CLINICAL TRIAL: NCT07272018
Title: Incidence and Clinical Significance of Maternal Hypotension After Labor Epidural Analgesia and Its Effects on Fetal Well-Being
Brief Title: Maternal and Fetal Clinical Significance of Hypotension Following Labor Epidural Analgesia
Status: Not yet recruiting | Type: Observational
Sponsor: The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Maxim Glebov, Staff Anesthesiologist in the Department of Anesthesiology, The Chaim Sheba Medical Center
Other Study IDs: SMC-2210-25
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Maternal Hypotension; Labor Epidural Analgesia; Fetal Heart Rate Abnormalities
Keywords: Labor Epidural Analgesia; Post-Epidural Hypotension; Maternal Hypotension; Fetal Heart Rate Abnormalities; Non-Reassuring Fetal Heart Rate; Obstetric Anesthesia
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laboring Participants Receiving Epidural Analgesia: This cohort includes adults in labor at Sheba Medical Center who choose to receive epidural analgesia for pain relief. All participants receive standard clinical care. Researchers will observe maternal blood pressure and fetal heart rate changes during the first 30 minutes after the epidural.
  Interventions: Other: Epidural Analgesia (Standard Clinical Care)

INTERVENTIONS:
Other: Epidural Analgesia (Standard Clinical Care) — Participants receive epidural analgesia for labor pain relief as part of routine clinical care at Sheba Medical Center. The epidural involves placement of an epidural catheter, a test dose, and a loading dose of local anesthetic according to hospital protocol. The study does not change how the epidural is performed. Researchers only observe maternal blood pressure and fetal heart rate after epidural placement.

SUMMARY:
The goal of this study is to learn how often blood pressure drops after an epidural for labor and how these drops may affect the parent and the baby. The study focuses on adults who give birth at term and choose to receive an epidural for pain relief.

The main questions the study aims to answer are:

How often does maternal blood pressure fall within 30 minutes after the epidural? When blood pressure falls, how often do participants need treatments such as fluids or medicines that raise blood pressure? Do changes in the baby's heart rate happen during this time, and do they need treatment? Are certain parent or labor factors linked to a higher chance of blood pressure drops? How often does an urgent cesarean delivery happen because of maternal low blood pressure or concerning fetal heart rate changes soon after the epidural?

Participants will not be asked to do anything different from usual care. Researchers will:

Review routine vital signs recorded before and after the epidural Review treatments given, such as IV fluids or blood-pressure-raising medicines Review the baby's heart-rate monitoring Record delivery information, including whether an urgent cesarean was needed This study does not change clinical care in any way. It uses information already collected during standard labor and delivery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* 37 weeks pregnant or more (term pregnancy)
* in labor and choose to receive an epidural for pain relief
* giving birth at Sheba Medical Center

Exclusion Criteria:

* patients with a heart condition that requires special blood pressure management
* medical conditions that prevent safe monitoring of blood pressure
* missing or incomplete medical record data needed for the study
* patient who do not receive an epidural during labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Laboring adults who receive epidural analgesia for pain relief at the labor and delivery unit of Sheba Medical Center, a large tertiary hospital in Israel. Participants represent people giving birth at term who choose epidural analgesia as part of their routine clinical care.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Absolute and relative number of patients with any MAP (mean arterial pressure) < 65 mmHg | First 30 minutes after epidural placement
  Hypotension after epidural placement

SECONDARY OUTCOMES:
Absolute and relative number of patients with any MAP (mean arterial pressure) < 60, 55 mmHg | First 30 minutes after epidural placement
  Hypotension after epidural placement
Absolute and relative number of patients with any SBP (systolic blood pressure) < 90, 85, 80 mmHg | First 30 minutes after epidural placement
  Hypotension after epidural placement
Incidence of postepidural hypotension defined as ≥20% MAP (mean arterial pressure) drop | First 30 minutes after epidural placement
  Hypotension after epidural placement
Absolute and relative number of patients with ≥20% SBP (systolic blood pressure) drop | First 30 minutes after epidural placement
  Hypotension after epidural placement
Time-to-treatment of Hypotension (minutes) | First 30 minutes after epidural placement
  The time interval between epidural placement and the treatment of hypotension by clinical staff
Area under a MAP of 65, 60, 55 mmHg [mmHg x min] | First 30 minutes after epidural placement
Absolute and relative number of patients with symptoms due to hypotension | First 30 minutes after epidural placement
  Weakness, lightheadedness, fainting, dizziness, nausea, vomiting
Absolute and relative number of patients with NRFHR (Non-reassuring fetal heart rate) | First 30 minutes after epidural placement
Absolute and relative number of patients who received fluid bolus | First 30 minutes after epidural placement
Absolute and relative number of patients who received vasopressor | First 30 minutes after epidural placement
  Phenylephrine, ephedrine
Absolute and relative numbers of patients who underwent urgent Cesarean section (Category 1 or 2 urgency) due to hypotension or NRFHR (non-reassuring fetal heart rate) | First 30 minutes after epidural placement

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ralston DH, Shnider SM. The fetal and neonatal effects of regional anesthesia in obstetrics. Anesthesiology. 1978 Jan;48(1):34-64. doi: 10.1097/00000542-197801000-00007. No abstract available. PMID 339784
- [Result] Ghidini A, Vanasche K, Cacace A, Cacace M, Fumagalli S, Locatelli A. Side effects from epidural analgesia in laboring women and risk of cesarean delivery. AJOG Glob Rep. 2023 Dec 12;4(1):100297. doi: 10.1016/j.xagr.2023.100297. eCollection 2024 Feb. PMID 38283322
- [Result] Paech MJ, Godkin R, Webster S. Complications of obstetric epidural analgesia and anaesthesia: a prospective analysis of 10,995 cases. Int J Obstet Anesth. 1998 Jan;7(1):5-11. doi: 10.1016/s0959-289x(98)80021-6. PMID 15321239
- [Result] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504